CLINICAL TRIAL: NCT02767999
Title: Resting State MRI Connectivity in Acute Ischemic Stroke: Serotonin Selective Reuptake Inhibitor (SSRI) in Enhancing Motor Recovery: a Placebo Controlled Study
Brief Title: Serotonin Selective Reuptake Inhibitor (SSRI) Effects on Cerebral Connectivity in Acute Ischemic Stroke
Acronym: RECONISE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC31/14/7388
Record Dates: First submitted 2016-05-06; First posted 2016-05-11 (Estimated); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Stroke
Keywords: Acute ischemic stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluoxetine (Experimental): One group will take a 20 mg of fluoxetine capsule per day from D0 to D90 and have fMRI
  Interventions: Drug: Fluoxetine; Radiation: fMRI
- Placebo (Placebo Comparator): The other group will take a cellulose placebo per day from D0 to D90 and have fMRI
  Interventions: Drug: Placebo; Radiation: fMRI

INTERVENTIONS:
Drug: Fluoxetine — 20 mg of fluoxetine capsule per day from D0 to D90
  Arms: Fluoxetine
Drug: Placebo — cellulose placebo per day from D0 to D90
  Arms: Placebo
Radiation: fMRI — functional resting state MRI

SUMMARY:
Fluoxetine action on cerebral connectivity changes in acute ischemic stroke patients

DETAILED DESCRIPTION:
In this placebo-controlled study, using functional resting state MRI, the investigators aim to investigate cerebral connectivity changes induced by fluoxetine given once a day for 90 days, in stroke patients with a moderate to severe motor deficit.

ELIGIBILITY:
Inclusion Criteria:

* First-ever ischemic stroke
* Cortical or subcortical stroke
* National Institute of Health Stroke Scale NIHSS>12 or motor NIHSS>6 at inclusion
* MRI-proved ischemic stroke

Exclusion Criteria:

* pregnant or breast-feeding women
* alcoholism
* ongoing Selective Serotonin Reuptake Inhibitor treatment or interruption < 1 month
* allergic reaction after SSRI administration
* MRI contraindication
* NIHSS>22
* Severe aphasia
* Coma

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Intracerebral connectivity in the motor network between fluoxetine and placebo group. | 90 days
  Intracerebral connectivity difference in the motor network, assessed by functional resting state MRI, between fluoxetine and placebo group after the treatment.

SECONDARY OUTCOMES:
Intracerebral connectivity in the motor network between good responders patients | 90 days
  Intracerebral connectivity difference in the motor network, assessed by functional resting state MRI, in fluoxetine and placebo good responders patients, defined by :
  * 8 points gain on the National Institute of Health Stroke Scale (NIHSS), assessed between D0 and D30 and between D0 and D90
  * or 2 points gain on the modified Rankin score (mRS) assessed between D0 and D30 and between D0 and D90.
Intracerebral connectivity in the motor network between non-responders patients | 90 days
  Intracerebral connectivity difference in the motor network, assessed by functional resting state MRI, in non-responders patients of fluoxetine and placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: François CHOLLET, MD PhD, Study Director — University Hospital, Toulouse
Locations (2):
- France (2):
  - Hôpital Pellegrin, Bordeaux
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No